CLINICAL TRIAL: NCT04361279
Title: A Phase III, Multicenter, Randomized, Double-blind Study Comparing the Efficacy and Safety of SIBP-02 (Rituximab Biosimilar) and Rituximab Combination With CHOP in Previously Untreated Subjects With CD20+ DLBCL
Brief Title: A Study Comparing SIBP-02 and Rituximab Combination With CHOP in Previously Untreated Subjects With CD20+ DLBCL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIBP-02-03
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIBP-02 (Experimental): Biological: SIBP-02, 375 mg/m2, intravenous infusion, administered on day1. Drug: Cyclophosphamide, 750 mg/m2, intravenous infusion, administered on day2. Drug: Doxorubicin Hydrochloride, 50 mg/m2, intravenous infusion, administered on day2.
  Drug: Vincristine Sulfate, 1.4 mg/m2, intravenous infusion, administered on day2.
  Drug: Prednisone Acetate Tablets, 100 mg, orally administered on day2-6, one time per day.
  Treatment cycle: 6 cycles, each cycle is 3 weeks.
  Interventions: Drug: SIBP-02
- Rituximab (Active Comparator): Biological: Rituximab, 375 mg/m2, intravenous infusion, administered on day1. Drug: Cyclophosphamide, 750 mg/m2, intravenous infusion, administered on day2. Drug: Doxorubicin Hydrochloride, 50 mg/m2, intravenous infusion, administered on day2.
  Drug: Vincristine Sulfate, 1.4 mg/m2, intravenous infusion, administered on day2.
  Drug: Prednisone Acetate Tablets, 100 mg, orally administered on day2-6, one time per day.
  Treatment cycle: 6 cycles, each cycle is 3 weeks.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: SIBP-02 — Injection，100mg/10ml
  Arms: SIBP-02
Drug: Rituximab — Injection，100mg/10ml
  Arms: Rituximab

SUMMARY:
This is a randomised, double-blind, positive drug parallel controlled equivalence clinical trial initiated at about 30 sites in China.

In the trial, it is planned to enroll 414 subjects, randomized to two treatment groups in a ratio of 1:1 to receive the test drug and the positive control.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old, male or female;
* Patients diagnosed as CD20-positive diffuse large B-cell lymphoma after histopathological or cytological examination and untreated;
* ECOG score ≤ 2 when enrolled;
* Echocardiography measured LVEF ≥ 50%;
* The laboratory indicators during the screening period shall meet the following criteria:

White blood cell count (WBC) ≥ 4.0 × 109/L or the lower limit of normal of the local laboratory; patients with bone marrow invasion, WBC ≥ 3.0 × 109/L; Absolute neutrophil count (ANC) ≥ 2.0 × 109/L or the lower limit of normal of the local laboratory; in the patients with bone marrow invasion, ANC ≥ 1.5 × 109/L; Hemoglobin (HB) ≥ 90 g/L; in the patients with bone marrow invasion, HB ≥ 80 g/L; Platelets (PLT) ≥ 100 × 109/L; in the patients with bone marrow invasion, PLT ≥ 75 × 109/L; Total bilirubin ≤ 1.5 times upper limit of normal (ULN); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; Alkaline phosphatase ≤ 1.5 × ULN in the patients without bone marrow invasion; Serum creatinine level ≤ 1.5 × ULN;

* Patients having at least one two-dimensional measurable lesion as the basis for evaluation: for intra-nodal lesions, ≥1.5 cm in the long diameter and ≥1.0 cm in the short diameter; for extra-nodal lesions, ≥1.0 cm in the long diameter;
* Patients with lymphoma International Prognostic Index (IPI) score of 0-2, with stage I to IV;
* Female at the childbearing age who show negative in the pregnancy test, and agree to take effective contraceptive measures during the study period and within 12 months after the last dose; male patients who agree to take effective contraceptive measures during the study period and within 3 months after the last dose;
* Patients with the expected survival period of greater than 6 months;
* Patients voluntary to sign the Informed Consent Form.

Exclusion Criteria:

* Patients with primary central nervous system lymphoma and secondary central nervous system invasion, gray zone lymphoma between Burkitt and DLBCL, gray zone lymphoma between DLBCL and HL, primary mediastinal DLBCL, primary exudative lymphoma, plasmablastic lymphoma, primary skin DLBCL, ALK-positive DLBCL or transformed lymphoma;
* Patients with double hit (BCL-2 and c-MYC gene rearrangement) or triple hit (BCL-2, BCL-6 and c-MYC gene rearrangement) diffuse large B-cell lymphoma diagnosed by the FISH test method; or patients with the pathological immunohistochemical test results as follows: BCL-2 ≥70% positive and c-MYC≥40% positive and tumor cells judged to be the source of germinal center according to Han's evaluation criteria but without exact FISH test result;
* Patients with history of malignant tumors other than cutaneous squamous cell carcinoma, cutaneous basal cell carcinoma and cervical carcinoma in situ within 5 years prior to enrollment;
* Patients with major surgery (excluding diagnostic surgery) within 2 months prior to enrollment;
* Patients treated for non-Hodgkin's lymphoma:

Chemotherapy and immunotherapy; Radiotherapy or local radiotherapy for DLBCL; Monoclonal antibody therapy (including Rituxan® and biosimilars of Rituxan®) Surgery (except biopsy);

* Patients previously receiving cytotoxic drugs or anti-CD20 antibodies to treat other diseases (e.g. rheumatoid arthritis);
* Patients receiving any monoclonal antibody within 3 months prior to enrollment;
* Patients who participated in other clinical trials and used other trial-related drugs within 3 months prior to enrollment;
* Those vaccinated within 1 month prior to enrollment;
* Those receiving hematopoietic cytokines, e.g. granulocyte colony-stimulating factor (G-CSF) within 2 weeks prior to enrollment;
* Those with the maximum dose of >100mg Prednisone Acetate Tablets or equivalent cortisols for more than 5 days for the purpose of controlling lymphoma, or with the daily dose of >30mg Prednisone Acetate Tablets or equivalent cortisols for more than 10 days for the other purposes. For the patients with daily dose of ≤30mg Prednisone Acetate Tablets or equivalent cortisols, there shall be written record on stable use of pre-randomization dose for at least 4 weeks;
* Patients with peripheral nervous system or central nervous system disorder;
* Patients with suspected active or latent tuberculosis;
* Patients with known uncontrolled active bacterial, viral, fungal, mycobacterial, parasitic or other infections (excluding nail bed fungal infection) or with any significant systemic infection event that requires intravenous antibiotic treatment or hospitalization (except for neoplastic fever) within 4 weeks prior to enrollment;
* HIV antibody positive;
* HCV antibody positive;
* HBV infection: (1) HBsAg positive, or (2) HBsAg negative, HBcAb positive and HBV DNA > 1 × 103
* Patients with complicated other diseases that might restrict the patients from participation in the clinical trial in the opinion of the investigator, including but not limited to:

Cardiovascular disease: congestive heart failure (NYHA Class III-IV), unstable angina, poorly controlled arrhythmias, poorly controlled hypertension or hypotension or myocardial infarction in the past 6 months; Severe mental illness; Gastric ulcer, intestinal infarction or gastrointestinal perforation (except for ones caused by primary disease); Pulmonary diseases (asthma, interstitial lung disease or severe obstructive pulmonary disease); Poorly controlled diabetes.

* Patients with contraindication to any drug in the CHOP chemotherapy regime;
* Patients with allergy constitution or known to be allergic to the active ingredient, excipient or rodent product or xenogeneic protein of any drug contained in this clinical trial (including the CHOP regime);
* Patients unsuitable for enrollment due to alcohol or drug abuse in the opinion of the investigator;
* Female in the pregnancy or breast-feeding period;
* Those unsuitable to participate in the clinical trial in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | After 6 cycles of treatment, each cycle is 3 weeks
  defined as the proportion of patients with Complete Response (CR) and Partial Response (PR) in accordance with the evaluation criteria of the International Working Group (IWG) Lymphoma Efficacy Evaluation System (2007)

CONTACTS AND LOCATIONS:
Overall Officials: Shanghai Institute Of Biological Products Co., Ltd, Study Director — SINOPHARM; The First Affiliated Hospital of College of Medicine, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided